CLINICAL TRIAL: NCT03172286
Title: Radiofrequency Technic's Impact on Perineal Postpartum Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-43; 2016-A01499-42 (Other: IDRCB)
Record Dates: First submitted 2017-03-30; First posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-03

CONDITIONS: Delivery; Injury
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Double blind study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient treated with fake radiofrequencer (Active Comparator)
  Interventions: Device: Radiofrequencer
- Patient treated with radiofrequencer (Experimental)
  Interventions: Device: Radiofrequencer

INTERVENTIONS:
Device: Radiofrequencer — Patients will be treated with a radiofrenquencer switched on or off depending on the attributed group after randomization

SUMMARY:
A study in the postpartum period reveals that among women who delivered vaginally and having perineal lesions, between 95 and 100% of them suffer from perineal pain (episiotomy, tears from 1st to 4th degree) to 24 hours of vaginal delivery; and between 60 and 91% 7 days after delivery.

Severe pain that is not taken into account can become chronic pain. It has physical and psychological consequences. It is therefore essential to prevent these risks in young mothers.

The main objective of this study is to assess the efficacy of radiofrequency treatment on perineal pain postpartum, after a vaginal delivery, instrumented or not, in patients with perineal lesions.

A double-blind randomized prospective single-center study will be conducted on patients delivering at Marseille's north hospital.

Women who gave birth to the North hospital site, with perineal lesions (tears, episiotomy) will be invited to enroll in the study.

Patients will be then randomized into two groups, one with radiofrequency treatment, the other without treatment with radiofrequency.

The duration of inclusion is provided over 6 months. Each topic will be followed over a period of 1 month. The total study duration is 7 months.

The expected results are a significant reduction in pain scores during the first days postpartum in women with perineal alteration caused by a vaginal delivery instrumented or not. Also an improvement in the quality of life of patients during the first days.

ELIGIBILITY:
Inclusion Criteria:

* Patients who naturaly delivered with ou without instruments such as Suction cup, spatulas, forceps
* Patients presenting perineal lesions

Exclusion Criteria:

* Patients who delivered through cesarean section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain score using analogical pain scale | 30 minutes
  Pain score will be assessed before and after the radiofrequencing cession

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Masreille, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bretelle F, Fabre C, Golka M, Pauly V, Roth B, Bechadergue V, Blanc J. Capacitive-resistive radiofrequency therapy to treat postpartum perineal pain: A randomized study. PLoS One. 2020 Apr 27;15(4):e0231869. doi: 10.1371/journal.pone.0231869. eCollection 2020. PMID 32339169